CLINICAL TRIAL: NCT03666117
Title: Prevalence of Hepatomegaly in Children and Adolescents With Type 1 Diabetes Mellitus Attending Assiut University Children Hospital
Brief Title: Prevalence of Hepatomegaly in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manar Khalifa Zohery Shazly, Seed pharmaceutical company street, Assiut University
Other Study IDs: 17100551
Record Dates: First submitted 2018-09-09; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Hepatomegaly
MeSH Terms: conditions — Hepatomegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: children and adolescents with type 1 diabetes

SUMMARY:
To assess the prevalence of hepatomegaly in children and adolescents with type 1 diabetes mellitus, and to find out it᾿s underlying etiology.

DETAILED DESCRIPTION:
Type 1 diabetes is a disorder of glucose metabolism that results from insulin deficiency secondary to autoimmune destruction of insulin-secreting β-cells. The prevalence of liver disease among diabetics is estimated to be between 17% and 100%(1).

Most of these data were obtained from studies of obese adults with non-insulin dependent diabetes(2). Data regarding frequency of aetiological causes of hepatomegaly in children and adolescent with type 1 diabetes mellitus are scanty even in international publication(2).

Diabetes mellitus (DM) is associated with various structural and functional liver abnormalities, including non-alcoholic fatty liver disease (NAFLD) and hepatic glycogenosis (HG)(3).

NAFLD represents the most common liver disease(3) and is more typically found in obese adults with T2DM secondary to insulin resistance, while (HG) is more common in patients with lower body mass index and pediatric patients(4).

HG involves pathological glycogen storage in hepatocytes and is characterized by hepatomegaly and a transient elevation in liver transaminases that is associated with poorly controlled DM, particularly type 1 diabetes (T1D)(5).

The differential diagnosis of hepatomegaly in diabetic patients must consider several other potential causes of liver damage, such as infection (e.g., viral hepatitis), metabolic disorders (e.g., α1-antitrypsin deficiency and Wilson's disease), obstruction, autoimmune liver disease, hemochromatosis and celiac disease(6).

Presence of hepatomegaly and/or hyperechogenic liver on ultrasound abdomen was an indication for further laboratory work up to investigate other possible liver pathologies .The screening work up included: HBV surface antigen, Anti-HCV antibody, serum immunoglobulins, anti-nuclear antibody, smooth muscle antibody qualitative test , serum ferritin, serum iron, transferring saturation, and total iron binding capacity, urine for organic acids and plasma for amino acids, to evaluate for possibility of viral hepatitis B and C, autoimmune liver disease, hemochromatosis, and metabolic disorder, respectively(7).

It was considered that the finding of hyperechogenic liver and/or hepatomegaly on ultrasound and negative screening work up for underlying liver disease as consistent with a likely diagnosis of hepatic glycogenosis or less likely fatty liver(8).

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 Diabetes mellitus diagnosed according to the diagnostic criteria of the American Diabetes Association 2011.

Exclusion Criteria:

- 1-Patients with type 2 diabetes mellitus 2-Patients with secondary diabetes 3-Patients with type 1 diabetes mellitus with other system affection rather than hepatic affection like ( Central nervous system, Respiratory, Renal, Cardiovascular).

4- Syndromic children. 5-Patients known to have liver disease prior to diagnosis of diabetes.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and adolescents
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Hepatomegaly in children and adolescents | 1 year
  the prevalence of different causes of hepatomegaly with type 1 diabetes mellitus .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut children hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
Time Frame: 1 year